CLINICAL TRIAL: NCT03665753
Title: Comparison of Intravenous Ketorolac 10, 20, and 30mg for Treating Renal Colic Pain in the Emergency Department: A Randomized Controlled Trial
Brief Title: Comparison of IV 10, 20, and 30mg for Renal Colic Pain in the ED
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hadi Mirfazaelian, Assistant Professor of Emergency Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9521307004
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pain; Renal Colic
MeSH Terms: conditions — Pain; Renal Colic | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: Dose escalation study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketorolac 10mg (Experimental): Subjects will be administered 10 mg of Ketorolac.
  Interventions: Drug: Ketorolac
- Ketorolac 20mg (Experimental): Subjects will be administered 20 mg of Ketorolac
  Interventions: Drug: Ketorolac
- Ketorolac 30mg (Experimental): As a part of standard care, subjects will be administered 30 mg of Ketorolac.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Subject will receive 10, 20, and 30mg of Ketorolac.

SUMMARY:
Hypothesis: Intravenous administration of Ketorolac 10 mg and 20 mg is as effective as 30 mg in treating renal colic pain in patients presenting to the emergency department

DETAILED DESCRIPTION:
Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that is widely used in the Emergency Department (ED). Because of the Ketorolac significant analgesic potency, it is usually used for moderate-to-severe pain. However, ketorolac has several side effects, of which gastrointestinal hemorrhage is most concerning. "Analgesic ceiling" is defined as the dose beyond which no additional analgesia can be achieved and on the other hand, more side effects might be encountered. Several studies suggested 10 mg as analgesic ceiling. Despite this, many recommendations are still advocating several folds higher doses (e.g. 30, 60 mg).

ELIGIBILITY:
Inclusion Criteria:

* Severe flank and abdominal pain which pertains to renal colic according to emergency physician's gestalt

Exclusion Criteria:

* Age >65
* Active Peptic Ulcer disease
* Acute Gastrointestinal Hemorrhage
* Known History of Renal or Hepatic insufficiency
* History of allergies to NSAIDs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Pain assessed with visual analogue scale (VAS) | 30 Minutes
  The visual analogue scale (VAS) will be used for the study. The VAS ranges from 0 (no pain) to 100 (very severe pain). The higher the pain scores the higher the pain severity.

SECONDARY OUTCOMES:
Pain assessed with visual analogue scale (VAS) | 15 Minutes
  The visual analogue scale (VAS) will be used for the study. The VAS ranges from 0 (no pain) to 100 (very severe pain). The higher the pain scores the higher the pain severity.
Pain assessed with visual analogue scale (VAS) | 45 Minutes
  The visual analogue scale (VAS) will be used for the study. The VAS ranges from 0 (no pain) to 100 (very severe pain). The higher the pain scores the higher the pain severity.
Pain assessed with visual analogue scale (VAS) | 60 Minutes
  The visual analogue scale (VAS) will be used for the study. The VAS ranges from 0 (no pain) to 100 (very severe pain). The higher the pain scores the higher the pain severity.
Adverse Effects | 60 Minutes
  Dizziness (Adverse Effect), Nausea (Adverse Effect), Vomiting (Adverse Effect), headache (Adverse Effect)

CONTACTS AND LOCATIONS:
Locations (1):
- IKCH, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eidinejad L, Bahreini M, Ahmadi A, Yazdchi M, Thiruganasambandamoorthy V, Mirfazaelian H. Comparison of intravenous ketorolac at three doses for treating renal colic in the emergency department: A noninferiority randomized controlled trial. Acad Emerg Med. 2021 Jul;28(7):768-775. doi: 10.1111/acem.14202. Epub 2021 Feb 17. PMID 33370510